CLINICAL TRIAL: NCT02858934
Title: Feasibility Study of Accelerated Preoperative Radiotherapy for Early Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andre Nazac (Other)
Responsible Party: Sponsor-Investigator, Andre Nazac, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUB-Preop-Breast
Record Dates: First submitted 2016-08-04; First posted 2016-08-08 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: Short preoperative tomotherapy; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preoperative tomotherapy (Experimental): This study is an open study investigating the effect on quality of life of a very short preoperative radiotherapy for early breast cancer, including approximately 24 women. Radiotherapy will be performed in 1 week and before the surgery in stead of following surgery.Preoperative radiotherapy has the advantage that the tumor is visible on imaging. This can result in smaller boost volumes. The surgery will follow shortly after termination of the radiotherapy, resulting in a very short treatment period.
  Interventions: Radiation: Tomotherapy

INTERVENTIONS:
Radiation: Tomotherapy — Dose prescription:
  Whole breast irradiation: 25 Gy in 5 daily fractions of 5 Gy Boost: 30 Gy in 5 daily fractions of 6 Gy The boost will be delivered as a simultaneous integrated boost (SIB).
  Target volumes:
  Clinical target volume (CTV) breast: defined by the soft tissue of the breast down to the pectoralis fascia, but excluding the skin and the underlying muscle, ribs, lung and heart.
  Gross tumor volume (GTV) boost: includes all gross tumor volume, as visible on computer tomography, mammography and/or magnetic resonance imaging (MRI). MRI imaging is preferentially performed in treatment position.
  CTV boost: includes the primary tumor, with a margin of 1.0 cm in all directions to encompass potential microscopic disease extension. The CTV boost excludes the skin, pectoralis muscle, ribs, lung and heart.
  Planning target volume (PTV): CTV plus a margin of 5 mm in all directions, but limited at 5 mm below the skin surface.

SUMMARY:
The standard treatment for women with a relatively small breast cancer without arguments for involvement of the axillary lymph nodes, is breast conserving surgery followed by radiotherapy of the whole breast, often with a complementary dose to the operated area (boost). A delay of 3-4 weeks after surgery is advisable for allowing wound healing before the start of radiotherapy. Historically, whole breast radiotherapy plus boost are delivered in 6-7 weeks. This treatment can be associated with temporary fatigue and decrease in quality of life. Randomized trials have shown that shorter schedules, delivering slightly more dose per day during 3 weeks, are equal to the long schedules. In an earlier clinical study, the investigators have tested such a short schedule and shown that it is equally safe and equally well tolerated as the conventional schemes. Other hospitals have examined (and still are examining) the safety and tolerance of even shorter schedules, delivering radiotherapy in 1 week.

This clinical study involves delivering radiotherapy in 1 week and before the surgery in stead of following surgery. In the postoperative setting, it is often debatable which volume should be included in the boost. Often boost-volumes remain large because of uncertainties in delineation. Preoperative radiotherapy has the advantage that the tumor is visible on imaging. This can result in smaller boost volumes. The surgery will follow shortly after termination of the radiotherapy, resulting in a very short treatment period.

This study is an open study investigating the effect on quality of life of a very short preoperative radiotherapy for early breast cancer.

DETAILED DESCRIPTION:
Women with early breast cancer are treated with breast conserving surgery (BCS) followed by whole breast irradiation (WBI) and a complementary dose to the lumpectomy cavity (boost). A delay of 3-4 weeks after surgery is advisable for allowing wound healing before the start of radiotherapy. Historically, WBI plus boost are delivered in 6-7 weeks. This treatment is associated with fatigue and a decreased quality of life. Randomized trials have shown that shorter hypofractionated schedules, delivering radiotherapy in 3 weeks, are equal to the long schedules. The investigators have shown that a hypofractionated tomotherapy with a simultaneous integrated boost is oncologically safe, well tolerated and has less impact on quality of life than the conventional schemes.

In the postoperative setting, it is often debatable which volume should be included in the boost. Surgical clips can help to decrease inter-observer variability, but often boost-volumes remain large because of uncertainties in delineation. Preoperative radiotherapy has the advantage that the gross tumor volume (GTV) is visible on imaging. This can result in smaller boost volumes.

The aim of this study is to investigate the feasibility of a short preoperative tomotherapy. The potential benefits are

* a decrease in overall treatment time
* a positive effect on quality of life
* a more precise target delineation
* profitable health economics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological diagnosis of unifocal invasive breast carcinoma, no special type (ductal carcinoma)
* Tumor Staging: cT1-2N0M0
* Luminal A or B
* Candidate for breast conserving surgery
* N0-status confirmed by lymph node cytology

Exclusion Criteria:

* Multifocal/multicentric disease
* Prior thoracic radiotherapy
* Pregnancy
* SBR3 grading
* Triple negative status which benefit neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Duration of the surgical procedure | from 2 to 8 days after the last radiotherapy session.
  Duration of the breast conserving surgery (lumpectomy + sentinel lymph node procedure)
Quantity of blood lost | from 2 to 8 days after the last radiotherapy session.
  Quantity of blood that has been lost during the breast conservation surgery, performed 2 to 8 days after the last radiotherapy session.
Dindo score | Week 6 after radiotherapy start
  Post operative morbidity assessment according to Dindo, Demartines et al.
Wound disruption (yes/no) | up to 30 days post operative
  Presence of wound disruption defined as skin dehiscence from any cause including seroma or hematoma.
Wound infection (yes/no) | up to 30 days post operative
  Presence of wound infection, defined as: purulent drainage, cellulitis, abscess or wound requiring drainage, debriding, and antibiotics associated with a clinical diagnosis of infection.
Number of adverse events | up to three months after radiotherapy start
  Acute radiation toxicity measure

SECONDARY OUTCOMES:
QLQ-C30 questionnaire | week 3 after radiotherapy start
  Assessment of the quality of life, according to the QLQC30 questionnaire
QLQ-C30 questionnaire | week 6 after radiotherapy start
  Assessment of the quality of life, according to the QLQC30 questionnaire
EORTC QLQ-BR23 questionnaire | week 3 after radiotherapy start
  Assessment of the quality of life, according to the EORTC BR23 questionnaire
EORTC QLQ-BR23 questionnaire | week 6 after radiotherapy start
  Assessment of the quality of life, according to the EORTC BR23 questionnaire
Number of adverse events | from three months after radiotherapy start till end of study (up to 1 years)
  Late toxicity measure
Local recurrence (yes/no) | up till the end of study (1 year)
  Local control: presence of local cancer recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Mark De Ridder, MD, Principal Investigator — CHU Brugmann/UZ Brussel
Locations (3):
- Belgium (3):
  - CHU Brugmann, Brussels
  - UZ Brussel, Brussels
  - AZ Sint Blasius, Dendermonde

REFERENCES:
- [Background] Senkus E, Kyriakides S, Ohno S, Penault-Llorca F, Poortmans P, Rutgers E, Zackrisson S, Cardoso F; ESMO Guidelines Committee. Primary breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v8-30. doi: 10.1093/annonc/mdv298. No abstract available. PMID 26314782
- [Background] Bartelink H, Horiot JC, Poortmans PM, Struikmans H, Van den Bogaert W, Fourquet A, Jager JJ, Hoogenraad WJ, Oei SB, Warlam-Rodenhuis CC, Pierart M, Collette L. Impact of a higher radiation dose on local control and survival in breast-conserving therapy of early breast cancer: 10-year results of the randomized boost versus no boost EORTC 22881-10882 trial. J Clin Oncol. 2007 Aug 1;25(22):3259-65. doi: 10.1200/JCO.2007.11.4991. Epub 2007 Jun 18. PMID 17577015
- [Background] Whelan TJ, Pignol JP, Levine MN, Julian JA, MacKenzie R, Parpia S, Shelley W, Grimard L, Bowen J, Lukka H, Perera F, Fyles A, Schneider K, Gulavita S, Freeman C. Long-term results of hypofractionated radiation therapy for breast cancer. N Engl J Med. 2010 Feb 11;362(6):513-20. doi: 10.1056/NEJMoa0906260. PMID 20147717
- [Background] Haviland JS, Owen JR, Dewar JA, Agrawal RK, Barrett J, Barrett-Lee PJ, Dobbs HJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Simmons S, Sydenham MA, Venables K, Bliss JM, Yarnold JR; START Trialists' Group. The UK Standardisation of Breast Radiotherapy (START) trials of radiotherapy hypofractionation for treatment of early breast cancer: 10-year follow-up results of two randomised controlled trials. Lancet Oncol. 2013 Oct;14(11):1086-1094. doi: 10.1016/S1470-2045(13)70386-3. Epub 2013 Sep 19. PMID 24055415
- [Background] Van Parijs H, Miedema G, Vinh-Hung V, Verbanck S, Adriaenssens N, Kerkhove D, Reynders T, Schuermans D, Leysen K, Hanon S, Van Camp G, Vincken W, Storme G, Verellen D, De Ridder M. Short course radiotherapy with simultaneous integrated boost for stage I-II breast cancer, early toxicities of a randomized clinical trial. Radiat Oncol. 2012 Jun 1;7:80. doi: 10.1186/1748-717X-7-80. PMID 22656865
- [Background] Versmessen H, Vinh-Hung V, Van Parijs H, Miedema G, Voordeckers M, Adriaenssens N, Storme G, De Ridder M. Health-related quality of life in survivors of stage I-II breast cancer: randomized trial of post-operative conventional radiotherapy and hypofractionated tomotherapy. BMC Cancer. 2012 Oct 25;12:495. doi: 10.1186/1471-2407-12-495. PMID 23098579
- [Background] van Mourik AM, Elkhuizen PH, Minkema D, Duppen JC; Dutch Young Boost Study Group; van Vliet-Vroegindeweij C. Multiinstitutional study on target volume delineation variation in breast radiotherapy in the presence of guidelines. Radiother Oncol. 2010 Mar;94(3):286-91. doi: 10.1016/j.radonc.2010.01.009. Epub 2010 Mar 2. PMID 20199818
- [Background] Kirby AN, Jena R, Harris EJ, Evans PM, Crowley C, Gregory DL, Coles CE. Tumour bed delineation for partial breast/breast boost radiotherapy: what is the optimal number of implanted markers? Radiother Oncol. 2013 Feb;106(2):231-5. doi: 10.1016/j.radonc.2013.02.003. Epub 2013 Mar 13. PMID 23490269
- [Background] Nichols EM, Dhople AA, Mohiuddin MM, Flannery TW, Yu CX, Regine WF. Comparative analysis of the post-lumpectomy target volume versus the use of pre-lumpectomy tumor volume for early-stage breast cancer: implications for the future. Int J Radiat Oncol Biol Phys. 2010 May 1;77(1):197-202. doi: 10.1016/j.ijrobp.2009.04.063. PMID 20394853
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542